CLINICAL TRIAL: NCT05627167
Title: Daytime Cyclic Enteral Nutrition Versus Standard Continuous Enteral Nutrition in the Intensive Care Unit: a Pilot Randomized Controlled Trial
Acronym: DC-SCENIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHM-2022/S03/04
Record Dates: First submitted 2022-11-16; First posted 2022-11-25 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Enteral Nutrition
Keywords: Intensive Care; Enteral nutrition; Organ Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Daytime Cyclic enteral nutrition (Experimental): Patients receive continuous isocaloric enteral feeding for 10 hours during the day (e.g. 08:00 to 18:00) via nasal or oro-gastric tube
  Interventions: Other: day time cyclic nutrition
- Continuous enteral nutrition (Active Comparator): Patients receive isocaloric enteral feeding continuously 24 hours a day via nasal or oro-gastric tube
  Interventions: Other: continuous nutrition

INTERVENTIONS:
Other: day time cyclic nutrition — Continuous isocaloric enteral feeding (1kcal/ml) with 4g of protein per 100 mL for 10 hours during the day (e.g. 08:00 to 18:00), via nasal or oro-gastric tube
  Arms: Daytime Cyclic enteral nutrition
Other: continuous nutrition — Isocaloric enteral feeding (1kcal/ml) with 4g of protein per 100ml, continuously 24 hours a day by nasal or oro-gastric tube
  Arms: Continuous enteral nutrition

SUMMARY:
Critical care patients experience systemic aggression, which may be the result of trauma, infection or other systemic inflammatory mechanisms. The initial phase of their illness is characterized by metabolic instability and increased catabolism. Nutrition goals in these patients are therefore, on the one hand, to provide sufficient caloric intake to cover energy expenditure while limiting the risks of inappropriate under-feeding, overfeeding- or re-feeding syndrome, and on the other hand, to meet the protein requirements linked to hypercatabolism. In the absence of contraindication, current recommandations state that an intensive care patient who cannot be fed orally, shoul receive continuous enteral nutrition over 24 hours by gastric tube within 48 hours of admission.

However, this 24-hour continuous nutrition method does not correspond to the physiological habit of the human species which includes a physiological nighttime fasting period.This fasting period induces a metabolic switch that regulates several pathways, including glycemic control, oxidative stressresistance and deoxyribonucleic acid (DNA) repair. Furthermore, it takes part un the synchronization of cellular circadian rhythms.

Investigator hypothetises that diurnal cyclic enteral nutrition may improve the prognosis of severe intensive care patients compared to continuous enteral nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years and over admitted to intensive care
* On invasive mechanical ventilation for less than 24 hours
* With an indication for exclusive enteral feeding by naso- or oro-gastric tube
* With an expected remaining duration of mechanical ventilation > 72 hours

Exclusion Criteria:

* Enteral feeding via tube already started
* Parenteral nutrition in progress or deemed necessary by the practitioner
* Active digestive haemorrhage as evidenced by fibroscopy or with need for transfusion
* Digestive surgery less than one month old
* History of mesenteric ischaemia
* History of gastrectomy, oesophagectomy, duodenopancreatectomy, bariatric surgery, short bowel syndrome
* Pregnant, lactating or parturient woman
* Body mass index < 18 kg/m2
* Person deprived of liberty by judicial or administrative decision, person under forced psychiatric care, person under legal protection (guardianship or curatorship)
* Lack of social security coverage
* Lack of consent or emergency procedure form
* Patient participating in another randomised clinical research study on feeding of resuscitation patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
Change of organ failures | Day 7
  Change is measured by evolution of the Sequential Organ Failure Assessment (SOFA) score at D7 compared with D0 in both groups

SECONDARY OUTCOMES:
Average daily caloric intake | Day 1 to Day 7
  Average daily caloric intake from enteral nutrition
Proportion of patients achieving > 80% of their recommended caloric intake at D7 | Day 7
Average daily protein intake | Day 1 to Day 7
  Average daily protein intake in grams
Vomiting | Day 1 to Day 10
  Number of days with vomiting (passage of nutrition into the mouth or the endoctracheal tube)
Diarrhea | Day 1 to Day 10
  Number of days with more than four episodes of liquid stools
Constipation | Day 1 to Day 10
  Number of stool free days
Intestinal ischemia | Day 1 to Day 10
  Number of patients suffering an episode of intestinal ischemia
Ventilator acquired pneumonia | Day 1 to Day 10
  Number of episodes of ventilator acquired pneumonias
Insulin consumption | Day 1 to Day 7
  Average insulin consumption expressed in international units per kg per day
Lactatemia | Day 1 to Day 7
  Mean lactatemia measured before the start of a new feeding cycle
Hypoglycemia | Day 1 to Day 7
  Number of days with at least one capillary blood glucose < 0.6 g/L
Ketonemia | Day 1 to Day 7
  Average capillary ketonemia measured in the morning before the start of a new feeding cycle
Bilirubin | Day 1 to Day 7
  Average total plasma bilirubin levels measured in the morning before the start of a new feeding cycle
Urea | Day 1 to Day 7
  Average plasma urea levels measured in the morning before the start of a new feeding cycle
Mortality | At Day 28
  Whether patient is alive or dead
Days without mechanical ventilation | Day 1 to Day 28
  Number of days without mechanical ventilation at D28
Days intubated | Day 1 to Day 28
  Number of days during the ICU stay where the patient received invasive mechanical ventilation

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU Angers, Angers
  - Centre Hospitalier Du Mans, Le Mans
  - CHRU Tours, Tours

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonnable request from the principal investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Callahan JC, Parot-Schinkel E, Asfar P, Ehrmann S, Tirot P, Guitton C. Impact of daily cyclic enteral nutrition versus standard continuous enteral nutrition in critically ill patients: a study protocol for a randomised controlled trial in three intensive care units in France (DC-SCENIC). BMJ Open. 2024 Jan 29;14(1):e080003. doi: 10.1136/bmjopen-2023-080003. PMID 38286683